CLINICAL TRIAL: NCT04048213
Title: The Becoming of Children With Doose Syndrome
Acronym: DOOSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Lille (Other); University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0058
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Doose Syndrome; Epileptic Syndromes; Learning Disabilities
Keywords: doose syndrome; Epileptic Syndromes; Learning Disabilities
MeSH Terms: conditions — Epilepsies, Myoclonic; Epileptic Syndromes; Learning Disabilities | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — questionnaire send to the parents

SUMMARY:
Doose syndrome is a rare epileptic syndrome that can lead to learning difficulties and a poor quality of life. The goal of this study is to evaluate the evolution of epilepsy and its consequences on cognitive development and learning issues in children with Doose syndrome.

DETAILED DESCRIPTION:
Doose syndrome is a rare epileptic syndrome beginning between ages two and five, characterized by myoclonic-astatic seizures which can be associated with myoclonic seizures, astatic seizures, absences and generalized tonic-clonic seizures. These seizures can be difficult to treat effectively and may lead to learning difficulties. During this study, parents of children with Doose syndrome will receive a questionnaire regarding learning disabilities, quality of life and epilepsy of their children.

ELIGIBILITY:
Inclusion Criteria:

* children with doose syndrome diagnosed between ages 1 and 6
* normal development until onset of seizures

Exclusion Criteria:

* unconfirmed diagnoses
* abnormal diagnoses
* abnormal psychomotor development before onset of seizures
* cerebral MRI abnormalities
* other child epileptic syndromes

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: During this study, parents of children with Doose syndrome will receive a questionnaire regarding learning disabilities, quality of life and epilepsy of their children. Children with doose syndrome diagnosed between ages 1 and 6 and with normal development until onset of seizures will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
disease effects on the learning ability of children with doose syndrome | day of inclusion
  disease effects on the learning ability of children with doose syndrome base on scholar informations

SECONDARY OUTCOMES:
Evolution of epilepsy in children with doose syndrome based on pathological symptoms | day of inclusion
  Evolution of epilepsy in children with doose syndrome based on pathological symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Nguyen, Pr, Principal Investigator — CHRU LILLE; Axel Lebas, MD, Principal Investigator — CHU Rouen
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No